CLINICAL TRIAL: NCT00388323
Title: Adipose Tissue Involvement in Alcohol-induced Liver Inflammation in Human : Study of Pro- and Anti-inflammatory Cytokines and ADIPOKINES..
Brief Title: Adipose Tissue Involvement in Alcohol-induced Liver Inflammation in Human
Acronym: RIHTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P 051041; AOR 05049
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-11

CONDITIONS: Alcoholic Hepatitis; Alcoholic Cirrhosis
Keywords: Alcohol; Hepatitis; Cirrhosis; Inflammation; Cytokines; ADIPOKINES; Adipose tissue
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Cirrhosis, Alcoholic; Hepatitis; Fibrosis; Inflammation | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: blood and biopsies

INTERVENTIONS:
Other: blood and biopsies — blood and biopsies

SUMMARY:
The histological characteristics of alcoholic liver disease (ALD) and non-alcoholic steatohepatitis (NASH) related to overweight and obesity suggest the presence of partly common physiopathological mechanisms. We reported that the ponderal overload was an independent risk factor of alcoholic cirrhosis. The adipose tissue was considered for a long time as a simple place of storage of fat. However, it is now recognized that the adipose tissue can secrete cytokines called ADIPOKINES.

The adipose tissue can secrete others cytokines such as TNF-alpha, IL6, IL10 and IL1-Ra. Increase in the production of the leptin and TNF-alpha by the adipose tissue after alcohol administration in the rat, as well as the role of leptin in inflammation and liver fibrogenesis in the murine model of chemical hepatotoxicity strongly suggest that activation of adipocytes by alcohol can explain the strong correlation observed between the body mass index (BMI) and the severity of ethanol-induced liver injury. Conversely, it was suggested in a murine model that the reduction in adiponectin production would sensitize the liver with the toxicity of alcohol. The PPAR alpha and gamma are the receptors which play a role both in inflammation and glucide and lipid metabolism. Taking into account the inhibiting role of PPAR alpha on the proliferation of the hepatic stellate cells, responsible for the fibrosis, the PPAR could also be implied in the relation between the overweight and the hepatic fibrosis in the alcoholic.

DETAILED DESCRIPTION:
The aim of this project is to demonstrate that ADIPOKINES, as well as the PPAR alpha and gamma are implied in the intensity of the steatosis and in the regulation of the inflammatory process and the hepatic fibrogenesis in alcoholic liver disease. In order to prove this hypothesis, we will study among patients having a ALD at various stages of histological severity: 1) the hepatic and subcutaneous abdominal adipose tissue expression of the PPAR alpha and PPAR gamma, 2) the hepatic and subcutaneous abdominal adipose tissue expression of the TNF alpha, the IL1Ra, the IL6 and the IL10, 3) the hepatic and subcutaneous abdominal adipose tissue expression of the ADIPOKINES (leptin, adiponectin, resistin), 4) the serum ADIPOKINES values, the cyanotic of the mRNA expression and of the serum ADIPOKINES values after 7 days of alcohol withdrawal 50 patients will be studied (25 having ALD without cirrhosis, with or without acute alcoholic hepatitis (AAH) and 25 having alcoholic cirrhosis with or without AAH). A part of liver biopsy will be frozen in a dry tube. The percutaneous adipose tissue will be obtained with a punction on the abdominal level at the time of inclusion of the patients having AAH and, for the second time, after 7 days of alcohol withdrawal, than will be frozen. The TNF alpha, the IL1Ra, the IL6, the IL10, the leptin, the adiponectin and the resistin expression as well as the hepatic and adipose tissue PPAR alpha and gamma will be evaluated by PCR in real time. The serum concentration of the ADIPOKINES (leptin, adiponectin, resistin) will be measured by ELISA or RIA.

If our hypothesis is true, severity of liver lesions (steatosis, AAH, fibrosis) could be positively correlated with the expression in the liver and the adipose tissue and / or the serum values of the anti-inflammatory cytokines and ADIPOKINES (TNF alpha, IL6, leptin, resistin) and negatively with the cytokines and ADIPOKINES which are potentially anti-inflammatory (IL1Ra, IL10, adiponectin). We also expect to find a negative correlation between the amount of hepatic and adipose tissue PPAR-alpha and PPAR-gamma mRNA and the severity of the liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Alcoholic patients of both sex aged from 18 to 75, hospitalized for alcoholic liver disease.
* HBs antigen negative, HIV negative, anti -VHC negative
* daily consumption exceeded 40-50 grams per day during the last year
* elevated AST level and liver biopsy during the hospitalisation Patients who signed the informed consent document
* patients affiliated to the national health insurance system

Exclusion Criteria:

* patients having another cause than alcohol for liver injury
* hepatocellular carcinoma or another developing cancer, severe associated pathology (cardiac disease, respiratory insufficiency, severe psychiatric problems), pancreatitis, infection, diabetes or a dyslipidemia
* patients treated with fibrates or other hypolipidaemic drugs, oral antidiabetics or insulin
* patients having hemostasis which does not permit the TRANSCOSTAL liver biopsy, platelet level <60 giga/l, or Quick test < 50 %, or (TCA higher than 1,5 times the time of the witness)
* patients refuse an adipose tissue biopsy
* patients treated with long-duration dose of clopidogrel (Plavix®)
* patients who significantly diminished alcohol consumption in comparison with the average consumption during the year preceding the inclusion
* patients not-affiliated to the national health insurance system

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Adipokines | at the inclusion and after one week
  To demonstrate that ADIPOKINES are implied in the intensity of the steatosis and in the regulation of the inflammatory process and the hepatic fibrogenesis in alcoholic liver disease.
PPAR α et γ | At the inclusion and after one week
  To demonstrate that the PPAR α et γ are implied in the intensity of the steatosis and in the regulation of the inflammatory process and the hepatic fibrogenesis in alcoholic liver disease.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel PERLEMUTER, MD, Principal Investigator — Hôpital Antoine Béclère - Clamart - FRANCE
Locations (1):
- Hôpital Antoine Béclère, Clamart, France

REFERENCES:
- [Derived] Voican CS, Njike-Nakseu M, Boujedidi H, Barri-Ova N, Bouchet-Delbos L, Agostini H, Maitre S, Prevot S, Cassard-Doulcier AM, Naveau S, Perlemuter G. Alcohol withdrawal alleviates adipose tissue inflammation in patients with alcoholic liver disease. Liver Int. 2015 Mar;35(3):967-78. doi: 10.1111/liv.12575. Epub 2014 Jun 3. PMID 24766056